CLINICAL TRIAL: NCT04467541
Title: A Randomized, Open, Phase I/II to Evaluate the Inactivated EV 71 Vaccine Safety in Healthy Adults Followed by Safety and Immunogenicity Administered in 2 Consecutive Doses, 1 Month Apart Among Child Aged 6 to 71 Months.
Brief Title: Safety & Immunogenicity of Enterovirus Type 71 Vaccine in Healthy Adults and Children 6-71months
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-19055
Record Dates: First submitted 2020-06-25; First posted 2020-07-13 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-06

CONDITIONS: Hand Foot & Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inactivated enterovirus type 71 vaccine (Experimental): Inactivated enterovirus type 71 vaccine safety in healthy adults followed by safety and immunogenicity administered in two consecutive doses, one-month apart among children aged 6 to 71 months
  Interventions: Biological: Inactivated Enterovirus Type 71 (EV71) Vaccine (Vero Cell)

INTERVENTIONS:
Biological: Inactivated Enterovirus Type 71 (EV71) Vaccine (Vero Cell) — Inactivated Enterovirus Type 71 (EV71) Vaccine safety in healthy adults followed by safety and immunogenicity administered in two consecutive doses, one-month apart among children aged 6 to 71 months
  Other Names: Inlive

SUMMARY:
1. Burden: Hand-foot-and-mouth disease (HFMD) characterized by skin rash in extremities, mouth ulcer and fever among <5 years children.Primarily caused by Enterovirus- predominantly human Enterovirus (EV) 71 and Coxsackie virus (CoxA). Several large epidemics have been reported worldwide.Large Asia-Pacific epidemic-in China in 2008, approximately 490,000 infections and 126 deaths of children. EV71 contributes severe and fatal cases e.g. encephalitis.A recent outbreak of HFMD in Bhubaneswar, Odisha in India indicates there is a chance of HFMD outbreaks in Bangladesh. However there is not much report of HFMD from Bangladesh.
2. Knowledge gap: EV71 is most commonly transmitted via close person-to-person contact. Since there is no known effective treatment for HFMD and as the causative virus is highly contagious, hand washing is the best defense for prevention. However, asymptomatic or mild nature of the infection leads to ineffectiveness of public health interventions like hand washing. Thus the symptomatic management remains the mainstay of treatment strategy for HFMD as of now. EV71 vaccine, an inactivated vaccine, developed by Sinovac Biotech Ltd has shown satisfactory safety and effectiveness through Phase III trials conducted in various regions of mainland China, This new vaccine has the potential to significantly reduce suffering and death from EV71 disease in China. However, it is not assessed on Bangladeshi child.
3. Relevance: Due to the absence of effective public health strategy and proper treatment, the development of an effective vaccine may be the best way to control EV71 infection.

DETAILED DESCRIPTION:
General objective:

1. To evaluate the safety of EV71 vaccine in adults and in children age 6-71 months
2. To evaluate the immunogenicity of the vaccine in children by assessing the neutralization antibody levels before immunization; then 7, 15, 30 days after the first inoculation; and also 7, 15, 30 days after the second inoculation.
3. To assess the incidence rate of adverse reactions/events

Specific objective: To find out:

1. Seroconversion rate of neutralization antibody on the day 30 after the whole-range immunization (i.e. after 2nd dose of vaccination);
2. Positive rate and Geometric Mean Titer of neutralization antibody on the day 30 after the whole-range immunization;
3. Seroconversion rate, positive rate and Geometric Mean Titer of serum neutralization antibody on the day 7, day 15, day 30 after the first inoculation;
4. Seroconversion rate,positive rate and Geometric Mean Titer of serum neutralization antibody on the day 7, day 15 after the second inoculation;
5. The incidence rate of adverse reactions & serious adverse events during the observation period of safety;
6. The incidence rate of adverse reactions 0-30 days after each inoculation of vaccine;
7. The incidence rate of adverse events 0-7 days after each inoculation of vaccine;

ELIGIBILITY:
Inclusion Criteria:

* Bangladeshi healthy adults 18-45yrs and children aged 6-71 months on the day of screening;
* Either sex;
* The participant /parents or guardian of the participant properly informed about the study and having signed the informed consent form (ICF);
* Participant/Parents' or guardian's availability for the entire period of the study and reachability by study staff for post-vaccination follow-up

Exclusion Criteria:

Exclusion Criteria for Inoculation of the First Dose:

Whether the participant should be enrolled should be judged according to the following criteria. The participant cannot participate in the study if any of the following circumstances exists:

1. Previous history of hand, foot and mouth disease;
2. Allergy history to vaccine or components of the vaccine, previous history of asthma, serious adverse effects of the vaccine such as urticaria, dyspnea, angioneurotic edema or stomachache, etc;
3. Congenital malformation or developmental disorder, genetic defect, serious malnutrition, etc;
4. Autoimmune disease or immunodeficiency or immunosuppression;
5. Severe neurological disorders (epilepsy, convulsion or tic) or family history of mental disease;
6. History of thyroidectomy, or asplenia or functional asplenia;
7. Severely malnourished children
8. Abnormal coagulation functions (such as coagulation factor deficiency, blood coagulation disease and blood platelet disorders) or obvious bruise or blood coagulation disorders diagnosed by the doctors;
9. Received immunosuppressant therapy, cytotoxic drug therapy and inhaled corticosteroid therapy (excluding the corticosteroid aerosol therapy for allergic rhinitis and surface corticosteroid therapy for acute non-complicated dermatitis) in the past 6 months;
10. Received blood products within 3 months before receiving the investigational vaccine;
11. Received other study drugs or vaccines within 30 days before receiving the investigational vaccine;
12. Received live attenuated vaccines within 14 days before receiving the investigational vaccine;
13. Received subunit or inactivated vaccines within 7 days before receiving the investigational vaccine;
14. Various acute diseases or acute exacerbation of chronic diseases within 7 days;
15. Fever before vaccine inoculation, axillary temperature >37.5°C;
16. Any other factors which are unsuitable for participation in the clinical trial as judged by the investigator.

Exclusion Criteria for Inoculation of the Second Dose of Vaccine:

1. Any serious adverse event related to the inoculation of the investigational product;
2. Hypersensitivity after vaccine inoculation (including urticaria/rash appeared within 30 minutes after inoculation);
3. Any confirmed or suspected autoimmune disease or immunodeficiency disease, including human immunodeficiency virus (HIV) infection;
4. If acute or newly onset chronic disease occurs during vaccine inoculation;
5. The investigator judged that other significant reactions occur (including serious pain, serious swelling, serious activity limitation, continuous hyperthermia, serious headache or other systemic or local reactions);
6. The patient develops acute disease when vaccine is inoculated (acute diseases means the moderate or severe disease with or without fever);
7. Axillary temperature >37.5°C when vaccine is inoculated;
8. The patient has received subunit inactivated vaccine within 7 days or live attenuated vaccines within 14 days.

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 430 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Neutralizing Antibody responses for evaluation of enterovirus 71( EV71) vaccines | before immunization, 7, 15, 30 days after the first inoculation, 7, 15, 30 days after the second inoculation
  Testing the neutralization antibody levels before immunization, 7, 15, 30 days after Ist inoculation, 7, 15, 30 days after the 2nd inoculation, calculate the positive seroconversion rate, the positive rate and geometric mean titre of neutralization antibody.
  Vaccine recipients will have greater increase in neutralization antibody titers (NT) after the first dose, without a further increase in NT after the second dose. The seroconversion rate will be increased after Ist & second inoculation
  Detection Method of the Anti-EV71 Neutralizing Antibody
  * Sample collection and processing
  * Serum will be examined to determine the potency of the neutralizing antibody
  * Treatment of the serum to be examined
  * Dilution of the serum to be examined and virus used for neutralization:
  * Serum and virus neutralizing and virus culture
  * Observation of the cytopathic change and judgment results

SECONDARY OUTCOMES:
Safety Outcome | After Ist vacctination (0 day) & 30 days after 2nd vaccination
  Solicited AE's (Local) e.g. Tenderness, Indurations, Redness, swelling Rash (Injection site), Pruritus with Grading & Solicited AE's (Systemic) e.g. Allergic Reaction, Fatigue, Asthenia, Dysphoria, Loss of Appetite Nausea, Vomiting, Diarrhea Fever (Axillary Temp)with Grading will be assessed.
  If any solicited or unsolicited AE's following vaccination in this study and will record adverse events at home in diary card.

CONTACTS AND LOCATIONS:
Overall Officials: Wasif Ali Khan, MBBS, MHS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh